CLINICAL TRIAL: NCT06658730
Title: Long-term Characterization of GORE® TAG® Conformable Thoracic Stent Graft With ACTIVE CONTROL System Performance
Acronym: TGR 23-02TA
Status: Recruiting | Type: Observational
Sponsor: W.L.Gore & Associates (Industry)
Responsible Party: Sponsor
Other Study IDs: TGR 23-02TA; TGR 23-02TA (Other: WL Gore)
Record Dates: First submitted 2024-10-16; First posted 2024-10-26 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Vascular Disease; Dissection; Dissection Aortic Aneurysm; Dissection of Aorta; Aneurysm Thoracic; Aneurysm Dissecting; Transection Aorta; Intramural Hematoma
Keywords: Endovascular; CTAG; Post-market Registry; Observational; Multi-regional; Real world data; Together Registry; Gore Together Registry; Gore Together Aortic Registry; Conformable Thoracic Stent Graft; TGR 23-02TA; TGR23-02TA; GORE TAG
MeSH Terms: conditions — Vascular Diseases; Aortic Dissection; Aortic Aneurysm, Thoracic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (2):
- Aneurysm/Other Isolated Lesion
  Interventions: Device: Endovascular
- Dissection
  Interventions: Device: Endovascular

INTERVENTIONS:
Device: Endovascular — TEVAR - thoracic endovascular aortic repair

SUMMARY:
An observational, prospective multi-regional post-market registry collecting mid- and long-term data to assess outcomes through ten years of follow-up for subjects treated with GORE® TAG® Conformable Thoracic Stent Graft with ACTIVE CONTROL System as a part of routine clinical practice. This post-market registry for the GORE® TAG® Conformable Thoracic Stent Graft with ACTIVE CONTROL System (CTAG w/AC) is intended to demonstrate that thoracic endovascular aortic repair (TEVAR) for lesions of the descending thoracic aorta continues to be a suitable treatment option for appropriately selected patients.

ELIGIBILITY:
Inclusion Criteria:

1. Patient or legally authorized representative (LAR) provides written authorization and/or consent per institution and geographical requirements.
2. Patient has been or is intended to be treated with an eligible registry device.*
3. Patient is age ≥ 18 years at time of informed consent signature.

   * The intent to treat a patient with a Gore product must be made prior to soliciting for possible registry participation. If pre-procedure consent is not feasible due to emergent situation, consent prior to the time of discharge for the index procedure is acceptable.

Exclusion Criteria:

1. Patient who is, at the time of consent, unlikely to be available for standard of care (SOC) follow-up visits as defined by the site's guidelines and procedures.
2. Patient with exclusion criteria required by local law.
3. Patient is currently enrolled in or plans to enroll in any concurrent investigational drug and/or investigational device study* within 12 months of Together Registry enrollment. Subjects cannot be enrolled in another Together Registry module protocol.

   * The term "study" does not apply to other observational registries or quality improvement projects. Collection of Registry Device performance from interventional studies may be permissible provided device application is not investigational and there are no novel requirements that alter follow-up conduct (i.e., protocol-mandated interventions).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The target registry population is patients who are treated with GORE® TAG® Conformable Thoracic Stent Graft with ACTIVE CONTROL at participating sites. This includes initial procedures and reinterventions (regardless of original intervention).
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2025-06-19 (Actual); Primary Completion 2038-08 (Estimated); Study Completion 2038-08 (Estimated)

PRIMARY OUTCOMES:
Deployment Technical Success | Index Procedure
  * Successful access, delivery, and accurate deployment of the device to the intended location, and retrieval of the delivery system.
  * The absence of any additional corrective procedure related to the device, procedure, or withdrawal of the delivery system. Events will not include interventions at the access site(s), lumbar drains to address spinal cord ischemia, or additional interventions to address non-treatment areas.
Lesion-related Mortality | From time of index procedure through 10 years of follow-up
  Death meeting at least one of the following characteristics:
  * Death within 30 days of the index procedure or following conversion to open repair.
  * Death within 30 days following a complication from a secondary procedure associated with the index lesion or registry device.
  * Any death where the treated disease / index lesion or registry device caused or significantly contributed to the death, including lesion-rupture, aortic-related complications, disease progression involving the index lesion.
Lesion Rupture (treated area) | Through 10 years post-procedure
  Rupture in the treated segment of the vessel (e.g., aorta or branch) verified with direct observation or CT / CTA scan.
Lesion Enlargement (treated area) | Through 10 years post-procedure
  An increase in maximum vessel (e.g., aorta or treated branch) diameter of > 5 mm in the region encompassed by the initial lesion as compared to baseline using orthogonal (i.e., perpendicular to the centerline) measurements on CT / CTA scans.
Endoleaks | Through 10 years post-procedure
  Perfusion of a treated lesion via:
  * Type I endoleak is defined as a sealing failure at one of the attachment zones of the graft to the vessel wall, whereby arterial flow perfuses the treated lesion via a perigraft channel:
    * Type Ia: Proximal aortic attachment zone
    * Type Ib: Distal aortic attachment zone
    * Type Ic: Distal attachment zone for branch component
  * Type II: Retrograde flow from native aortic branch arteries
  * Type III endoleak: Component disconnection or fabric disruption resulting in arterial flow into the perigraft space
    * Type IIIa: Attachment of aortic components (aortic-aortic)
    * Type IIIb: Fabric tear or disruption
    * Type IIIc: Attachment of aortic component-side-branch or side-branch-side-branch
  * Type IV: Late endoleak due to flow through porous fabric
  * Type V/Endotension: Aneurysm sac enlargement > 5 mm with no imaging evidence of an endoleak
  * Indeterminate: Endoleak is identified, but source cannot be ascertained
Device Migration | Through 10 years post-procedure
  Longitudinal movement of all or part of the device for a distance ≥ 10 mm, as confirmed by CTA scan, relative to anatomical landmarks and device positioning at the first post-operative CTA scan.
Loss of aortic / branch patency | Through 10 years post-procedure
  No flow or contrast detected through the implanted aortic and/or branch component (for branched devices) confirmed with imaging and/or direct observation.
Stroke (All, Serious, Non-Serious) | Through 10 years post-procedure
  Stroke is the acute onset of symptoms consistent with focal or multifocal Central Nervous System (CNS) injury caused by vascular blockage resulting in ischemia or vascular rupture resulting in hemorrhage, that:
  * Persists for > 24 hours or until death -or-
  * Symptoms lasting < 24 hours, with pathology or neuroimaging confirmation of CNS infarction
Paraplegia (within 30 days of index procedure) | Within 30 days of index procedure
  New onset spinal cord injury rendering a subject non-ambulatory within 30 days of the index procedure
Paraparesis (within 30 days of index procedure) | Within 30 days of index procedure
  New onset spinal cord injury causing a minor motor deficit of the lower extremities within 30 days of the index procedure
New onset renal failure (within 30 days of index procedure) | Within 30 days of index procedure
  New onset sustained renal failure identified within 30 days of the index procedure, combined with requiring dialysis for > 4 weeks
Renal function deterioration | Within 30 days of index procedure
  New onset of a decrease in eGFR > 30% following treatment when compared to baseline eGFR.
Device integrity events (e.g., fracture, kinking, compression) | Through 10 years post-procedure
  Defined as any of the following:
  * Wire fractures, including stents, hooks, or barbs
  * Stent kinking: Narrowing of the stent graft associated with demonstrable angulation in any of the stent components, with demonstrable flow
  * Disruption/tears in the graft component of the stent graft Stent compression or invagination: Transient or permanent stent-graft collapse following complete device deployment, resulting in an overall reduction in the vessel luminal diameter
Reintervention | Through 10 years post-procedure
  Additional surgical or interventional procedure related to the treated disease / index lesion, the registry device, or to the treatment / procedure.
  This may include surgical or interventional treatment for endoleaks, access site(s) complications, disease progression (including interventions to address issues related to non-treated area of the index lesion, such as bare stent implantation to address bowel ischemia associated with aortic dissection), spinal drains for Spinal Cord Injury (SCI) management, or conversion to open surgery.

SECONDARY OUTCOMES:
Access-related complications | Intra-operatively
  Complications associated with the access sites used during treatment that may include pseudoaneurysm, hematoma, thrombosis, or complications associated with percutaneous closure devices.
Transient Ischemic Attack (TIA) | Through 10 years post-procedure
  Transient focal neurological signs or symptoms (lasting <24 h) presumed to be due to focal brain ischemia but without evidence of acute infarction by neuroimaging or pathology (or in the absence of imaging)
New Dissection | Through 10 years post-procedure
  A new arterial tear either caused by a stent graft, natural disease progression or iatrogenic injury from endovascular manipulation. This can include the propagation, or extension, of a previous dissection that was not present at the time of initial presentation.
False Lumen Status - treated segment | Through 10 years post-procedure
  Status of the false lumen within the segment of the aorta initially treated with an endovascular stent graft:
  * Patent: Flow present throughout the entire aortic false lumen (absence of thrombus) on arterial-phase or delayed contrast-enhanced imaging.
  * Partial thrombosis: Thrombus or clot within the aortic false lumen but with a residual patent ﬂow channel on arterial-phase or delayed contrast-enhanced imaging.
  * Complete thrombosis: Complete thrombosis of the aortic false lumen on arterial- and delayed-phase imaging.
False Lumen Status - untreated segment | Through 10 years post-procedure
  Status of the false lumen outside of the segment of the aorta initially treated with an endovascular stent graft:
  * Patent: Flow present throughout the entire aortic false lumen (absence of thrombus) on arterial-phase or delayed contrast-enhanced imaging.
  * Partial thrombosis: Thrombus or clot within the aortic false lumen but with a residual patent ﬂow channel on arterial-phase or delayed contrast-enhanced imaging.
  * Complete thrombosis: Complete thrombosis of the aortic false lumen on arterial- and delayed-phase imaging.
False Lumen Perfusion | Through 10 years post-procedure
  Flow into the false lumen via:
  * Type IA entry ﬂow: ﬂow between the proximal endograft and aortic wall allowing systemic pressure antegrade ﬂow into the primary entry tear and proximal false lumen
  * Type IB entry ﬂow: distal entry tear adjacent to endograft due to septal fenestration or a new intimal tear at the distal aspect of the stent graft (dSINE) allowing systemic pressure direct ﬂow into the false lumen
  * Type II entry ﬂow: retrograde entry ﬂow through arch vessel branches (innominate, carotid, subclavian) or thoracic bronchial and intercostal arteries into the false lumen
  * Type R entry ﬂow: antegrade entry ﬂow from the true lumen into the false lumen through distal branch fenestrations (uncovered intercostal arteries, visceral or renal arteries, lumbar arteries, iliac branches) or septal fenestrations (excluding SINE)

OTHER OUTCOMES:
Health Economic and Quality of Life Data Analysis | Through 10 years post-procedure
  A Health Economic analysis is planned as part of the clinical registry. Initial analyses will only involve data that is collected within the registry CRFs. The objective of the Health Economic analysis is to understand the short- and long-term healthcare resource use and costs of the treatment(s) studied during the period of the clinical registry. Quality of life will also be evaluated at some sites within the Europe, Middle East and Africa (EMEA) regions and Asia-Pacific (APAC) regions, as applicable, using a standard survey.

CONTACTS AND LOCATIONS:
Overall Officials: Ali Azizzadeh, M.D., Principal Investigator — Cedars-Sinai Medical Center; Timothy Resch, Principal Investigator — Univ. of CPH - Denmark; Kazuo Shimamura, Principal Investigator — Osaka University Hospital - Japan
Locations (10):
- United States (3):
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Indiana University School of Medicine, Indianapolis, Indiana
  - Duke University, Durham, North Carolina
- Rigshospitalet, Copenhagen, Denmark
- Centre Hospitalier Universitaire Strasbourg, Strasbourg, France
- Germany (2):
  - Universitatsmedizin Frankfurt, Frankfurt
  - Regensburg University Hospital, Regensburg
- Laiko General Hospital of Athens, Athens, Greece
- Hospital Universitari de Bellvitge, Barcelona, Spain
- Uppsala University, Uppsala, Sweden

IPD SHARING:
Plan to Share IPD: No